CLINICAL TRIAL: NCT05950425
Title: The Effect of Aspiration Education Given by Different Methods on the Anxiety and Hopelessness Level of Mothers Whose Child is in Intensive Care: A Randomized Controlled Trial
Brief Title: Aspiration Training Given With Different Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Semra Kose, Asisstant Proffessor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEUSKose2
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Aspiration; Pediatric Intensive Care Unit
Keywords: Educational Methods; Child; Mother; Anxiety; Hopelessness
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental I group (video training + standard training) (Experimental): This group will be trained with the aspiration training video shot by the researcher on the model. The video content will include the introduction of the materials used in the aspiration application, how to maintain sterility, the position to be given to the child during aspiration, and the sterile aspiration on the model. After obtaining the consent of the mothers in Experiment I group who participated in the study and were assigned by randomization method, they will be taken to the day room of the service and the training video will be watched on the computer. After the end of the video, if they have any questions, they will be answered and they will be taken to their child's intensive care room after wearing the equipment (bonnet, shoe covers, apron, mask) necessary for the standard education and providing hand hygiene.
  Interventions: Other: Aspiration training
- Experimental II group (education booklet training + standard training) (Experimental): Aspiration training will be given to this group with a picture training booklet. The training booklet includes the purpose of aspiration, the materials to be used, the position to be given to the child during aspiration, the preservation of sterility, and the application of aspiration. Expert opinion will be taken for the training booklet to be used. After obtaining the consent of the mothers in the Experimental II group, who participated in the study and were assigned with the randomization method, they will be taken to the day room of the service and aspiration training will be given with a picture training booklet. After the training, the questions of the mothers will be answered. At the end of the illustrated training booklet training, mothers will be put in the necessary equipment (bone cap, shoe covers, apron, mask) for standard practice training and hand hygiene will be provided and they will be taken to the intensive care environment to their children's rooms.
  Interventions: Other: Aspiration training
- Control group (No Intervention): The routine standard training given to this group in aspiration training will be used. In this training, one-to-one telling and showing are available. After obtaining the consent of the mothers in the control group who participated in the study and were assigned by randomization method, the necessary equipment (bone cap, shoe covers, apron, mask) will be put on and hand hygiene will be provided and they will be taken to the intensive care unit. After the mother is taken to the room where the child is staying, the equipment and apparatus connected to her child (monitor, infusion pump, NG probe, foley catheter, endotracheal tube, tracheostomy, etc.) will be introduced, equipment used in the treatment process of her child (mechanical ventilator, oxygen valve, aspirator, ambu, aspiration). probe, etc.) will be introduced and physical contact with the child will be supported and ensured.

INTERVENTIONS:
Other: Aspiration training — Pre-test application; All mothers whose children are hospitalized in the PICU will be filled in the questionnaires after verbally expressing and signing the informed consent before being admitted to the intensive care unit and starting the education.
  In practice; The mother of the child who is planned to be discharged from the intensive care unit is given training a week before. Aspiration training will be given to the Experimental I group with the video method, and to the Experimental II group with the picture training booklet method. The materials of these trainings will be given to the mothers and they will be asked to look after them when they come to the next care.
  Final test application; scales will be filled in the mother on the day of the child's discharge.
  Arms: Experimental I group (video training + standard training); Experimental II group (education booklet training + standard training)

SUMMARY:
Parents whose children are in intensive care have to cope with many stressors in terms of psychological, physical, economic and social aspects. Especially during the discharge process, many reasons such as the fact that their children have a chronic disease, need for care, parents do not know how to provide the care their children need, the lack of professional health care teams provided by home care in our country, and therefore the care of the children is covered by the families, increase the anxiety levels of the parents. It increases the frequency of hospitalization of children or prolongs the length of stay in the intensive care unit, as appropriate care cannot be provided. In addition, frequent hospitalizations can cause damage to family dynamics. It has been determined that as the child grows, the difficulties experienced in the care of the child, the financial difficulties increase, the worries about the future and the constant relationship with the experts increase the stress of the parents and the stress is in parallel with the level of hopelessness. This is the factor that reinforces the anxiety and hopelessness in the daily life of parents. The fact that mothers whose children are in intensive care do not know the materials used, the procedures performed, the steps of the procedure, and what situations they will encounter at home may increase their stress-anxiety and hopelessness levels. Today, with the rapid development of technology, the use of educational technologies on the basis of learning and teaching has become widespread in health care education in the field of health, as in every field. It is important to address more than one sense organ in order for the education in the field of health to be more effective. Therefore, it is important to reduce the anxiety and hopelessness levels of the parents, to increase the self-confidence of the parents, to see general (physiological and psychological) improvements in children, and to reduce health costs with the training given to mothers with different education methods. The aim of this study is to determine the effect of aspiration training given by different methods on the level of anxiety and hopelessness of mothers whose children are in intensive care.

DETAILED DESCRIPTION:
Pediatric Intensive Care Units (PICUs) are units that have the necessary technical equipment and materials in order to maintain the life, care and treatment of children aged 1 month to 18 years who are in need of medical care, with one or more organ failure, and to prevent possible complications. It differs from other pediatric services where professional nursing care is provided with close follow-up and treatment.

Diseases admitted to the PICU include sepsis, status epilepticus, Central Nervous System infection, hepatic coma, animal bites/stings, traumas, intracranial hemorrhage, suffocation, electric shock, and meningococcemia, with the most common pulmonary infection being the most common. Hospitalization of the child for reasons such as illness, accident or injury can cause significant changes in almost the entire life of the family and cause anxiety. The fact that children's illnesses and injuries require hospitalization in intensive care makes the stress more traumatic. Being a member of the intensive care team, nurses, being aware of the stress sources of the parents whose children are hospitalized in the PICU and knowing their reactions can help them to cope with this situation.

There are no professional home care teams in our country to provide home care for children with special needs dependent on medical devices. Therefore, the care needs of these patients are met by their families after discharge. During the rehabilitation process of children with special care needs, the family may have to perform the duties of health professionals such as administering medication or oxygen therapy in general, performing routine maintenance and replacing tracheostomy tubes, maintaining airway patency, maintaining and replacing nasogastric tubes. After discharge, doing these cares takes a large part of the parents' attention, time and costs. It can cause stress, anxiety, and fear. Another factor affecting the anxiety levels of families after discharge is that they do not feel adequately equipped and educated for their children's care at home (aspiration, mechanical ventilator support, etc.), they do not know what to do in an emergency, they do not receive home health care services or they cannot reach enough. These are situations such as fear of being harmed at home because they think that their children are more sensitive and prone to getting sick than other children.

There are factors that prevent parents with special needs children from coping with the negative emotions they experience while raising their children, and one of them is their hope-level cognition and sensory status. This situation may be the factors that turn his daily life into anxiety and reinforce his hopelessness. Parents need to receive some training from nurses in order to fully care for their children who need special care. It is necessary to inform parents about the development of their child's self-care skills, to increase their ability to manage stress and to solve problems, and to encourage parents with the educational content prepared by determining the functions that the child needs care for.

ELIGIBILITY:
Inclusion Criteria:

* Having aspiration application in the treatment of the child
* Parent's ability to read and speak Turkish
* Parent's willingness to participate in the study
* Parent over 18 years of age
* The child has reached the discharge stage
* The mother has not done aspiration before
* Hospitalization of the child in the intensive care unit between the working dates

Exclusion Criteria:

* Variation of the child's health status during education
* Parent has a mental illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only mothers will be included in the study as more mothers take care of children in need of special care in Turkish society.
Enrollment: 84 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form: | 1st day
  The questionnaire prepared by the researcher considering the literature consists of 22 questions. This form consists of three parts: 10 questions about the child, 7 questions about the parent and family characteristics, and 5 questions about the mother's anxiety.

SECONDARY OUTCOMES:
The Beck Hopelessness Scale: | 1st and 8th day
  The scale was prepared by Beck et al. in 1974 with Heimber's anxiety about the future scale and with the help of clinicians. Seber (1991) translated it into Turkish in his associate professorship thesis, and then Seber, Dilbaz, Kaptanoğlu, and Tekin, (1993) and Durak (1994) conducted reliability studies. It is a measurement tool prepared to be applied to adolescents and adults in order to measure the negative expectations of the individual for the future. It is a scale consisting of 20 items and scored between 0-1. The score range is 0-20. High scores; indicates hopelessness and low indicates hope. A score of 0-3 indicates no or minimal hopelessness, a score of 4-8 indicates a low level of hopelessness, a score of 9-14 indicates moderate hopelessness, and a score of 15 and above indicates a high level of hopelessness.

OTHER OUTCOMES:
State Anxiety Inventory | 1st and 8th day
  The State-Anxiety Inventory was developed by Speilberger et al. (1980) to measure state and trait anxiety. The scale was adapted to Turkish by Öner and Le Comte (1983), and validity and reliability studies were conducted. The state and trait anxiety inventory consists of two separate sections and 40 items. The State Anxiety Inventory (STAI-1 / DKE) determines how a person feels at a known moment and under certain conditions. The lowest score to be obtained from the DCI is 20, and the highest is 80. Score between <0-40 according to the scale score: "No anxiety"; A score of 41-60: "Mild anxiety"; A score of 61 and above is evaluated as "severe anxiety"> (Öner & Le Compte, 1983).

CONTACTS AND LOCATIONS:
Overall Officials: Semra KÖSE, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan Üniversity, Meram, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The decision to share the study results will be made during the study period or when it is concluded

REFERENCES:
- [Background] Ağdaş D. (2008) Opinions of mothers of children hospitalized in the pediatric service of Cumhuriyet University Hospital regarding patient admission procedures and their expectations from nurses (Master's Thesis). Cumhuriyet University Institute of Health Sciences, Sivas. Ak, B. (2018). Child and nursing approach with chronic and life-threatening/fatal disease. Z. Conk, Z. Başbakkal, H. Bal Yılmaz, B. Bolışık (Ed.) in Pediatric Nursing (pp. 901- 936). Ankara: Academician Bookstore. Akşit S. & Cimete G. (2001) The effect of nursing care applied to mothers on the anxiety level of mothers when the child is admitted to the intensive care unit. C. U. Journal of the School of Nursing. 5(2): 25-36. Asatekin Yazgu, H. (2022). The Effect of Perceived Social Support on Anxiety and Anxiety Levels of Mothers with Their Baby in the Neonatal Intensive Care Unit [Unpublished master's thesis]. Istanbul University. Ayar, G., Şahin, S. , Yazıcı, M. U. , Coşkun, R. , Yakut, H. İ. & Demirel, F. (2015). Evaluation of Home Care Services in Pediatric Patients. Turkish Journal of Pediatrics, 9 (1) , 12-17 Aykanat Girgin, B. & Balcı, S. (2015). Home Care Needs of Physically Handicapped Children and Their Families. Gumushane University Journal of Health Sciences, 4 (2), 305-317 Biket, A. P., & Tönük, S. (2012). Examining the history of pediatric intensive care units and the current situation in Turkey with examples. Sigma, 4, 64-76. Bolışık, B. Z., Akçay Didişen, N., & Yavuz, B. (2014). Investigation of Use of Wet Wipes in Care of Mothers with Inpatient Children in Children's Hospital. Journal of Ege University Faculty of Nursing, 30(1), 91-100. Caicedo, C. (2014). Families With Special Needs Children. Journal of the American Psychiatric Nurses Association, 20(6), 398-407. https://doi.org/10.1177/1078390314561326